CLINICAL TRIAL: NCT06794749
Title: Investigation of the Effect of Action Observation Therapy Applied With Telerehabilitation Method on Upper Extremity Functions, Daily Living Activities and Quality of Life in Chronic Stroke Patients
Brief Title: Action Observation Therapy in Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Mustafa Kavak, Lecturer, MsC, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Karabuk-01
Record Dates: First submitted 2025-01-16; First posted 2025-01-27 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action Observation Therapy (Experimental): Patients received action observation therapy in addition to general physiotherapy via telerehabilitation method, 3 days a week for 5 weeks.
  Interventions: Other: Action Observation Therapy
- Control (Active Comparator): Patients received general physiotherapy in addition to face-to-face action observation treatment 3 days per week for 5 weeks.
  Interventions: Other: Control

INTERVENTIONS:
Other: Action Observation Therapy — Patients received general physiotherapy in addition to action observation therapy (AOT) via telerehabilitation method for 5 weeks, 3 days a week. AOT was applied to patients as a single session per day and lasted 30 minutes. General physiotherapy session was applied face to face for 45 minutes.
  Arms: Action Observation Therapy
Other: Control — Patients received general physiotherapy in addition to action observation therapy (AOT) via face-to-face telerehabilitation method for 5 weeks, 3 days a week. AOT was applied to patients as a single session per day and lasted 30 minutes. General physiotherapy session was applied face-to-face for 45 minutes.
  Arms: Control

SUMMARY:
Functional impairment in the upper extremities is one of the most common sequelae in stroke patients. It significantly limits the patients' grasping-releasing functions and, consequently, their activities of daily living (ADL), such as eating - drinking, dressing, and self-care. Action Observation Training (AOT), performed by observing simple actions frequently used in ADL and then imitating the observed actions, reduces interhemispheric inhibition and allows the elimination of impairments in upper extremity motor function and relearning of functions in chronic stroke patients. This study aims to investigate the effects of telerehabilitation and face-to-face AOT application on upper extremity functions, activities of daily living, and quality of life in chronic stroke patients and to question whether there are differences between the short- and long-term effects of these two AOT applications.

DETAILED DESCRIPTION:
Stroke is defined as a neurological picture caused by focal damage to the central nervous system due to vascular problems such as cerebral infarction or intracerebral or subarachnoid hemorrhage.

Functional impairment in the upper extremities is one of the most common sequelae in stroke patients. It significantly limits the patients' grasping-releasing functions and, consequently, their activities of daily living (ADL), such as eating - drinking, dressing, and self-care.

Action Observation Therapy (AOT), which is performed by observing simple actions frequently used in ADL and then imitating the observed actions, is a rehabilitation approach used in recent years to improve upper limb functions in the rehabilitation of stroke and various neurological diseases. It is stated that AOT reduces interhemispheric inhibition and allows the elimination of impairments in motor function and relearning of functions.

Telerehabilitation is the remote delivery of rehabilitation services through telecommunication technology. Telerehabilitation provides important advantages, such as difficulty transferring the patient to the health center, where the rehabilitation process takes a long time, travel time, and travel costs in stroke patients.

In the literature review, no study was found comparing the effect of the AOT with the telerehabilitation method and face-to-face application on the patient's upper extremity functions, activities of daily living, and quality of life in the rehabilitation of patients with chronic stroke. In addition, to our knowledge, there is no study examining the long-term effects of AOT, which has been the subject of a limited number of studies.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age,
* Diagnosis of left hemiparetic stroke,
* Having passed between 6-36 months since the onset of stroke,
* Being in stage 4 or 5 of the hand and stage 4, 5 or 6 of the upper extremity according to Brunnstrom staging,
* Being able to sit on a chair for 30 minutes without support (patients who scored 20 or more points in total from the Trunk Impairment Scale),
* Scoring 24 or more points from the Mini Mental Test

Exclusion Criteria:

* Not volunteering to participate in the study,
* Having spasticity (level 3 and 4 according to the Modified Ashworth Scale) that prevents grasping and releasing an object,
* Having contracture in any of the upper extremity joints on the affected side,
* Having a serious neglect disorder (scoring 21 and above on the Catherine Bergego Scale),
* Having cooperation, adaptation and behavioral disorders during the application of the tests used to obtain the data,
* Having mental impairment that prevents communication and receiving basic commands (scoring less than 24 on the Mini Mental Test)
* Having additional neurological and/or orthopedic problems that may affect motor performance and sitting balance
* Having advanced vision and hearing problems (if any, these problems have not been corrected with assistive devices such as glasses, lenses, hearing aids, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Spasticity | Baseline
  Spasticity will assessed using the Modified Ashworth Scale. As the score increases, spasticity increases. The minimum score for this scale is 1 and the maximum score is 5.
Stage of hemiplegia | Baseline
  "Brunnstrom Hemiplegia Recovery Staging" will be used to determine the hemiplegic stage of the patients. This scale is scored between 1 and 6. As the score increases, the patient improves.
Motor function | Baseline, five week later (after intervention), 3 months later
  The "Fugl-Meyer Upper Extremity Motor Assessment Scale" will be used to evaluate upper extremity motor functions. This scale ranges from 0 to 66 points. As the score increases, motor function improves.
Dominant side | Baseline
  The "Edinburgh Hand Preference Test" will be used to determine the dominant side used by the patient in daily life.
Trunk Impairment | Baseline
  "Trunk Impairment Scale" will be used to evaluate trunk impairment in stroke patients. The maximum score that can be obtained from the scale is 23 points. A low score indicates poor performance, a high score indicates good performance
Upper extremity function | Baseline, five week later (after intervention), 3 months later
  Evaluation of upper extremity functions (hand-arm) and motor speed will be done with the "Nine-Hole Peg Test". Function decreases as the time spent for the test increases.
Functional Independence | Baseline, five week later (after intervention), 3 months later
  Evaluation of upper extremity functions will be done with the "Nine-Hole Peg Test". Function decreases as the time spent on the test increases.
Cognitif Function | Baseline
  Mini Mental Test will be used to evaluate cognitive functions. In the evaluation, 24-30 points indicate that cognitive functions are normal, 18-23 points indicate mild cognitive impairment, and 17 points and below indicate that cognitive status is severely affected.
Neglect | Baseline
  The Catherine Bergego Scale will be used to assess the impact of unilateral neglect after stroke on activities of daily living. 1-10 indicates mild neglect, 11-20 indicates moderate neglect, and 21-30 indicates severe neglect.
Life Quality | Baseline, five week later (after intervention), 3 months later
  The Stroke Specific Quality of Life Scale will be used to assess the quality of life of individuals with stroke. The higher the total score, the better the quality of life of the individual with stroke. This scale is scored between 49-245.As the score increases, the quality of life increases.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa KAVAK, MsC, Principal Investigator — Karabuk University
Locations (1):
- Mustafa KAVAK, Karabük, Karabük Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Friberg H, Lundberg D, Nilstun T. [Ethical views on resuscitation. Formal guidelines for do-not-resuscitate orders in Sweden]. Lakartidningen. 1994 Oct 19;91(42):3787-9. No abstract available. Swedish. PMID 7996947
- [Result] Cortes-Gallegos V, Sojo Aranda I, Gio Pelaez RM. Disturbing the light-darkness pattern reduces circulating testosterone in healthy men. Arch Androl. 1998 Mar-Apr;40(2):129-32. doi: 10.3109/01485019808987935. PMID 9507745
- See also: Research study — https://www.annexpublishers.com/articles/JNND/7104-The-Comparison-between-the-Effect-of-Action.pdf